CLINICAL TRIAL: NCT01560455
Title: The European Bifurcation Coronary Study; A Randomised Comparison Of Provisional T-Stenting Versus A Systematic Two Stent Strategy In Large Calibre True Bifurcations
Brief Title: European Bifurcation Club Trial - Two-stent Versus One-stent Technique for Large Bifurcation Lesions
Acronym: EBC TWO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Sussex County Hospital (Other)
Collaborators: Terumo Corporation (Industry)
Responsible Party: Principal Investigator, David Hildick-Smith, Consultant Cardiologist, Royal Sussex County Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EBC TWO
Record Dates: First submitted 2011-09-16; First posted 2012-03-22 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Disease
Keywords: stent; bifurcation; coronary
MeSH Terms: conditions — Coronary Disease | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single stent (Active Comparator): single stent
  Interventions: Device: single stent
- dual stent (Active Comparator): dual stent (culotte)
  Interventions: Device: two stent

INTERVENTIONS:
Device: single stent — single stent
  Other Names: Terumo Nobori stent
  Arms: single stent
Device: two stent — culotte
  Other Names: Terumo Nobori stent
  Arms: dual stent

SUMMARY:
This study will examine use of two-stent versus one-stent techniques for patients with large calibre bifurcation lesions including significant side branch disease.

DETAILED DESCRIPTION:
Treatment of bifurcation coronary lesions remains a difficult area, in which best practice is yet to be established. Prior to the era of drug-eluting stents, the limited data which existed suggested that a strategy of stenting the main vessel, with balloon angioplasty alone of the side-branch if required was superior to stenting both vessels.

Randomised trials of "all-comer" bifurcation lesions have now established that there is no advantage to systematic dual drug-eluting stent strategies. However, these trials included patients with no disease in the side branch, and small side branch vessels.

Expert consensus suggests that "large" bifurcations with significant ostial side branch disease still merit a systematic total lesion coverage stent technique. This trial therefore is designed to assess the hypothesis that large true bifurcations with significant side branch ostial disease are more successfully treated with a systematic culotte technique than with the provisional T approach.

ELIGIBILITY:
Inclusion Criteria:

* "True" coronary bifurcation lesion (i.e. >50% lesion in both main vessel and side branch) requiring revascularisation
* Main vessel ≥ 2.5mm diameter (visual inspection)
* Side branch ≥ 2.5mm diameter (visual inspection)
* Side branch ostial lesion ≥5mm length
* Patient ≥18 years old
* Females of childbearing potential: -ve pregnancy test

Exclusion Criteria:

* Acute ST elevation myocardial infarction
* Cardiogenic shock
* Left main stem lesion of haemodynamic significance
* Chronic total occlusion of either vessel
* Additional Type C lesions requiring PCI
* Either bifurcation vessel not suitable for stenting
* Platelet count ≤50 x 109/mm3
* Left ventricular ejection fraction ≤20%
* Patient life expectancy less than 12 months
* Known allergies to aspirin, clopidogrel, heparin, stainless steel, intravenous contrast (severe), or stent drug elutant
* Participation in another investigational drug or device study
* Patient unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Composite primary endpoint (Death, MI, TVR) | 12 months
  Death Myocardial infarction Target Vessel Revascularisation

SECONDARY OUTCOMES:
Stent thrombosis | 12 months
  Stent thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Sussex Cardiac Centre, Brighton, East Sussex, United Kingdom

REFERENCES:
- [Derived] Arunothayaraj S, Behan MW, Lefevre T, Lassen JF, Chieffo A, Stankovic G, Burzotta F, Pan M, Ferenc M, Hovasse T, Spence MS, Brunel P, Cotton JM, Cockburn J, Carrie D, Baumbach A, Maeng M, Louvard Y, Hildick-Smith D. Stepwise provisional versus systematic culotte for stenting of true coronary bifurcation lesions: five-year follow-up of the multicentre randomised EBC TWO Trial. EuroIntervention. 2023 May 16;19(4):e297-304. doi: 10.4244/EIJ-D-23-00211. Online ahead of print. PMID 37946522
- [Derived] Hildick-Smith D, Behan MW, Lassen JF, Chieffo A, Lefevre T, Stankovic G, Burzotta F, Pan M, Ferenc M, Bennett L, Hovasse T, Spence MJ, Oldroyd K, Brunel P, Carrie D, Baumbach A, Maeng M, Skipper N, Louvard Y. The EBC TWO Study (European Bifurcation Coronary TWO): A Randomized Comparison of Provisional T-Stenting Versus a Systematic 2 Stent Culotte Strategy in Large Caliber True Bifurcations. Circ Cardiovasc Interv. 2016 Sep;9(9):e003643. doi: 10.1161/CIRCINTERVENTIONS.115.003643. PMID 27578839